CLINICAL TRIAL: NCT01953068
Title: Executive Reaction Time Test in Assessment of Cognitive Dysfunction After Aortic Valve Procedures
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Kati Järvelä, Kati järvelä, MD, PhD, Tampere University Hospital
Other Study IDs: R13043
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Neurobehavioral Manifestations
Keywords: POCD; Executive Reaction Time Test; Aortic valve surgery; Cognitive functions; Transcatheter Aortic Valve Implantation
MeSH Terms: conditions — Neurobehavioral Manifestations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Up to 50% of patients undergoing surgical aortic valve operation suffer from some level of post-operative cognitive dysfunction (POCD). Frontal lobes of the brain, where executive functions are located, are highly susceptible to trauma caused by possible blood malperfusion to these areas of the brain during surgery. Conventional and established neuropsychological test methods are poor in distinguishing these kinds of trauma, as they are isolated, structured tests that do not require multitasking and processing of multiple stimuli at the same time.

The phase 1 goal of this study is to employ an experimental Executive reaction time (RT) test to see if this method could improve objective detection of subtle brain dysfunction assumed to underlie persistent cognitive, somatic, and affective complaints reported by patients who have undergone electic aortic valve replacement (AVR) surgery. Phase 2 of the study will concentrate on patients undergoing transcatheter aortic valve implantation (TAVI).

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective aortic valve stenosis surgery (phase 1) or transcatheter aortic valve implantation (phase 2)

Exclusion Criteria:

* Previous neurological or psychiatric disorder.
* Significant visual problem
* Problems with upper arm/hand use

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective aortic valve replacement (AVR) and transcatheter aortic valve implantation (TAVI) patients at Tampere University Hospital Heart Center
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Executive Reaction Time Test response speed | 6 months

SECONDARY OUTCOMES:
Executive Reaction Time Test: error% of answers | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonne Liimatainen, MD, Principal Investigator — Tampere University Hospital; Kaisa Hartikainen, Professor, Study Director — Behavioral Neurology Research Unit, Pirkanmaa Hospital District; Arvi Yli-Hankala, Professor, Study Director — Tampere University Hospital; Kati Järvelä, MD, PhD, Principal Investigator — Tampere University Hospital Heart Center
Locations (2):
- Finland (2):
  - Tampere University Hospital Heart Center, Tampere, Pirkanmaa
  - Tampere University Hospital, Tampere

REFERENCES:
- [Derived] Liimatainen J, Perakyla J, Jarvela K, Sisto T, Yli-Hankala A, Hartikainen KM. Improved cognitive flexibility after aortic valve replacement surgery. Interact Cardiovasc Thorac Surg. 2016 Oct;23(4):630-6. doi: 10.1093/icvts/ivw170. Epub 2016 May 30. PMID 27245618